CLINICAL TRIAL: NCT01065220
Title: The Influence of Sex Steroid Hormones on Serotonin Transporter Binding in the Human Brain Investigated by Positron Emission Tomography
Brief Title: Sex Steroids and the Serotonin Transporter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AP13214ONB
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Transsexualism
Keywords: Serotonin Transporter; Hormone therapy; Gender Dysphoria; Transsexualism
MeSH Terms: conditions — Transsexualism; Gender Dysphoria | interventions — testosterone undecanoate; Lynestrenol; Cyproterone Acetate; Estradiol; 5-alpha Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hormone treatment for MtF (Experimental): * cyproterone acetate
  * estradiol
  * alpha-5-reductase-inhibitor
  Interventions: Drug: Cyproterone Acetate; Drug: Estradiol; Drug: 5-alpha reductase inhibitor
- hormone treatment for FtM (Experimental): * testosterone undecanoate
  * lynestrenol
  Interventions: Drug: Testolactone undecanoate; Drug: Lynestrenol

INTERVENTIONS:
Drug: Testolactone undecanoate — 4ml i.m.
  Other Names: Nebido®
  Arms: hormone treatment for FtM
Drug: Lynestrenol — 2/day
  Other Names: Orgametril®
  Arms: hormone treatment for FtM
Drug: Cyproterone Acetate — 50mg per day
  Other Names: Androcur®
  Arms: hormone treatment for MtF
Drug: Estradiol — 100 microgram TTS twice a week
  Other Names: Estradot®
  Arms: hormone treatment for MtF
Drug: 5-alpha reductase inhibitor — 1mg daily
  Other Names: Finasterid®
  Arms: hormone treatment for MtF

SUMMARY:
The aim of this study is to prove the influence of the sex steroid hormones estrogen, progesterone and testosterone on the serotonin transporter (5-HTT) binding using positron emission tomography (PET) and the selective radioligand [11C]DASB. Specifically, the 5-HTT binding will be quantified before and after hormone therapy underwent by 10 male-to-female (MtF) and 10 female-to-male (FtM) transsexuals urging for hormone treatment. The high-level, long-term administration of opsite sex steroid hormones in transsexuals provide the unique opportunity to investigate the influence of sex steroid hormones on the serotonergic system. Since the serotonin transporter serves as a primary target molecule for antidepressant treatment, the results of the study will be of benefit for the assessment of the clinical relevance of estrogen and testosterone as modulatory and neuroactive agents.

ELIGIBILITY:
Inclusion Criteria:

* somatic health
* no previous sex hormone medication
* willingness to sign the written informed consent

Exclusion Criteria:

* severe diseases
* steroid hormone treatment within 6 months prior inclusion
* treatment with psychotropic agents such as selective serotonin reuptake inhibitors (SSRIs)
* any implant or stainless steel graft
* positive urine pregnancy test in women at the screening visit at each PET day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
change in serotonin-transporter binding potential (BP) in predefined brain regions, measured by Positron Emission Tomography | 5 months
  The serotonin-transporter BP will be assessed in a 90 min. dynamic PET measurement session at three timepoints: before start of hormonal therapy, after four weeks of hormonal therapy, and after 4 months of hormonal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, MD A/Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kranz GS, Wadsak W, Kaufmann U, Savli M, Baldinger P, Gryglewski G, Haeusler D, Spies M, Mitterhauser M, Kasper S, Lanzenberger R. High-Dose Testosterone Treatment Increases Serotonin Transporter Binding in Transgender People. Biol Psychiatry. 2015 Oct 15;78(8):525-33. doi: 10.1016/j.biopsych.2014.09.010. Epub 2014 Sep 23. PMID 25497691